CLINICAL TRIAL: NCT06626217
Title: Comparison of Perfusion Index Monitoring Using a Smartwatch and a Pulse Oximeter
Acronym: PIWATCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NVT_02_2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Perfusion Index
Keywords: Pulse oximetry; Perfusion index; Finger replantation; Smartwatch
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Interventional prospective single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of perfusion index monitoring using a smartwatch and a pulse oximeter (Experimental): Placing the finger pulse oximeter sensor on the left middle finger and placing the Massimo Watch W1 on the volunteer's left wrist (2 cm from the processus styloideus). Four interventions subsequently follow (Resting condition, Movement artifacts and Circulation constriction, Physical Exercise).
  Interventions: Other: Resting conditions; Other: Movement artifacts; Other: Circulation constriction; Other: Physical exercise

INTERVENTIONS:
Other: Resting conditions — The volunteers hand is at rest and Perfusion index readings are taken for six minutes from pulse oximeter and smartwatch
Other: Movement artifacts — The volunteer periodically spreads his/her fingers and clenches them into a fist, and Perfusion index readings are taken for six minutes from pulse oximeter and smartwatch.
Other: Circulation constriction — The volunteers arm is constricted using a cuff to measure non-invasive blood pressure. The perfusion index value is monitored during the time of cuff pressure and cuff release. The measurement is followed by a 4-minute pause to allow the vascular supply to stabilize. The measurement is repeated three times.
Other: Physical exercise — The volunteer is seated on the exercise bike, rests his forearms on the handlebars and is instructed not to move his arms. The volunteer's heart rate is controlled to increase to 120 beats per minute. For five minutes, the perfusion index is recorded from a pulse oximeter and smartwatch.

SUMMARY:
The aim of the study is to experimentally compare measured perfusion index values between smartwatch and a medical grade pulse oximeter in healthy subjects at rest and with and without motion artifacts and during exercise.

DETAILED DESCRIPTION:
Perfusion index (PI) is one of the many vital signs monitored to assess the clinical status of a patient. PI is determined from the pulsatile part of the plethysmographic curve, with typical values measured on the fingers ranging from 0.02% to 20%. Although PI is a relatively newly measured parameter, it has already found application in many areas of clinical medicine. For example, continuous measurement of the perfusion index has been used to monitor changes in finger blood flow after finger replantation (surgical reattachment of the finger to the patient's body). As the ability to monitor the perfusion index begins to become part of the monitored parameters of smartwatches, this new feature could be used in situations where the use of finger sensors is not appropriate. However, no comparison of perfusion index measurements between smartwatch and pulse oximeter has been made to date.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult Volunteer

Exclusion Criteria:

* Post-traumatic upper limb conditions affecting finger or arm perfusion
* Injuries or diseases of the skin of the fingers and arm
* Any acute phase of any disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of measured perfusion index values between pulse oximeter and smartwatch during different interventions. | 1 hour
  The comparison of measured perfusion index values between pulse oximeter and smartwatch during different interventions (Resting conditions, Movement artifacts, Circulation costriction and Physical exercise) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Study Chair — Czech Technical University, Fac. of Biomedical Engineering

IPD SHARING:
Plan to Share IPD: Yes
The measured data will be shared publicly in the data repository on web page: https://ventilation.fbmi.cvut.cz/data/
Supporting Information: SAP
Time Frame: Unlimited from the time of processing complete measured data
Access Criteria: Publicly available to everyone
URL: https://ventilation.fbmi.cvut.cz/data/